CLINICAL TRIAL: NCT07301528
Title: Comparative Effects of Erector Spinae Plane and Quadratus Lumborum Blocks on Postoperative Pain and Analgesic Requirement in Pediatric Appendectomy: A Prospective Randomized Controlled Trial
Brief Title: Comparison of ESP and QL Blocks for Postoperative Pain in Pediatric Appendectomy (ESP-QLB)
Acronym: ESP-QLB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeycan Kahya (Other)
Responsible Party: Sponsor-Investigator, Zeycan Kahya, Medicine of Doctor, Kutahya City Hospital
Organization: Kutahya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KSBU-ESPQL-2026
Record Dates: First submitted 2025-11-16; First posted 2025-12-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Quadratus Lumborum Nerve Block; Erector Spinae Block
Keywords: Erector Spinae Plane Block; Quadratus Lumborum Block; Regional Anesthesia; Pediatric Appendectomy; Postoperative Pain; Ultrasound-Guided Nerve Blocks; Analgesic Requirement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel intervention arms: ultrasound-guided Erector Spinae Plane block or ultrasound-guided Quadratus Lumborum block, both performed under general anesthesia before surgical incision.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB Block (Experimental): Ultrasound-guided transmuscular QL block using 0.25% bupivacaine (0.5 mL/kg) before surgical incision.
  Interventions: Drug: Quadratus Lumborum Block (QLB)
- ESP Block (Active Comparator): Ultrasound-guided ESP block at the L1 level using 0.25% bupivacaine (0.5 mL/kg) before surgical incision.
  Interventions: Drug: Erector Spinae Plane Block

INTERVENTIONS:
Drug: Quadratus Lumborum Block (QLB) — Ultrasound-guided transmuscular QL block performed under general anesthesia using 0.25% bupivacaine (0.5 mL/kg) before surgical incision.
  Arms: QLB Block
Drug: Erector Spinae Plane Block — Ultrasound-guided ESP block at the L1 level under general anesthesia using 0.25% bupivacaine (0.5 mL/kg) before surgical incision.
  Arms: ESP Block

SUMMARY:
This prospective randomized controlled clinical trial aims to compare the analgesic effectiveness of the Erector Spinae Plane (ESP) block and the Quadratus Lumborum (QL) block in pediatric patients undergoing appendectomy. Both regional anesthesia techniques have been shown to reduce opioid requirements and improve postoperative recovery in children; however, there is limited evidence directly comparing their efficacy. In this study, eligible participants will be randomly assigned to receive either an ESP or a QL block in addition to standard general anesthesia before surgical incision. Postoperative outcomes will include pain scores, total opioid consumption, time to first analgesic requirement, mobilization time, parental satisfaction, length of hospital stay, block-related complications and block performance time. The findings are expected to guide clinicians in selecting the most effective regional anesthesia technique for postoperative pain control in pediatric appendectomy.

DETAILED DESCRIPTION:
Appendectomy is one of the most common emergency surgical procedures in children, and effective postoperative analgesia plays a key role in patient comfort, early mobilization, and reduced opioid exposure. Regional anesthesia techniques have gained increasing importance in pediatric anesthesia due to their opioid-sparing effect and favorable safety profile. Among these techniques, the Erector Spinae Plane (ESP) block and the Quadratus Lumborum (QL) block have shown promising results; however, there is a lack of high-quality randomized controlled trials directly comparing their clinical efficacy in pediatric appendectomy.

This study will prospectively enroll pediatric patients between 3 and 13 years of age who are scheduled to undergo appendectomy. After obtaining informed parental consent, participants will be randomly allocated to either the ESP block group or the QL block group. All blocks will be performed under ultrasound guidance using 0.25% bupivacaine at a dose of 0.5 mL/kg following the induction of general anesthesia. Standardized postoperative analgesia protocols will be applied to all participants.

Pain scores will be measured at predefined time points using a validated pediatric pain scale. Secondary outcomes will include total opioid consumption during the first 24 hours, the time to first rescue analgesic requirement, mobilization time, length of hospital stay, parental satisfaction scores, and any block-related complications. Patient data will be collected by trained investigators who will be blinded to group allocation.

The goal of this trial is to determine whether ESP or QL block provides superior postoperative pain control and recovery in pediatric appendectomy. The results may contribute to evidence-based recommendations for regional anesthesia selection in pediatric surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3-13 years
* Diagnosis of acute appendicitis requiring appendectomy
* ASA physical status I-II
* Planned general anesthesia with intraoperative regional block (ESP or QL block)
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Refusal of regional block by family or anesthesia team
* Coagulopathy or anticoagulant medication use
* Local infection at the block injection site
* Known allergy or contraindication to local anesthetics
* Neurological or neuromuscular disorders
* Cognitive impairment preventing postoperative pain assessment
* Conversion to open surgery
* Intraoperative complications requiring deviation from study protocol

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score | Pain scores will be assessed at 1, 6, 12, and 24 postoperative hours.
  Pain intensity will be evaluated at rest using the Oucher Pain Rating Scale. Higher scores indicate greater pain.

SECONDARY OUTCOMES:
Total Analgesic Consumption | Recorded during the first 24 hours after surgery
  Total dose of analgesic medications (NSAIDs and/or non-opioid analgesics) administered within the first 24 hours after surgery will be recorded. Higher values indicate greater analgesic requirement.
Time to First Analgesic Requirement | From the end of surgery until the first documented analgesic requirement, assessed up to 24 hours postoperatively
  Time interval between the end of surgery and the first administration of rescue analgesia will be recorded in minutes. Longer intervals indicate better analgesic effectiveness.
Time to Mobilization | From the end of surgery until the first successful ambulation with or without assistance, assessed up to 24 hours postoperatively
  Time from the end of surgery until the patient is able to ambulate with assistance or independently will be recorded in minutes. Shorter time indicates faster functional recovery.
Length of Hospital Stay | From the end of surgery until hospital discharge, typically within 24-48 hours.
  Duration of hospitalization will be recorded from admission to discharge and expressed in hours. Longer duration indicates delayed recovery.
Parents' Postoperative Pain Measure (PPPM) | Assessed at 1, 6, 12, and 24 hours postoperatively
  Postoperative pain will be evaluated by parents using the Parents' Postoperative Pain Measure (PPPM). Higher scores indicate greater pain intensity.
Block-Related Complications | From block performance until the end of surgery and during the first 24 hours postoperatively
  ny adverse events potentially related to the regional block (e.g., local hematoma or bruising, infection at the injection site, neurological symptoms, or suspected local anesthetic systemic toxicity) will be recorded as present or absent.
Block performance time | During block performance, prior to surgical incision
  Block performance time was defined as the time (in seconds) from the initial placement of the ultrasound probe on the skin to the completion of local anesthetic injection. The duration was recorded by an independent observer using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Camgöz, Principal Investigator — Kutahya Health Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Kutahya City Hospital Anesthesia and Reanimation Department, Kütahya, Kütahya
  - Kutahya City Hospital, Kütahya

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  Individual participant data (IPD) underlying the published results (de-identified) will be available upon reasonable request for research purposes.
  Supporting Materials:
  Statistical analysis code and study protocol will be available upon request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 6 months after publication of the study results and continuing for 2 years.
Access Criteria: Researchers must submit a methodologically sound proposal. Data will be shared after approval by the principal investigator. Data will be transferred in de-identified form only.